CLINICAL TRIAL: NCT01387074
Title: A Prospective, Non-interventional, Observational Study of Botox® Treatment for Patients With Upper Limb Adult Spasticity
Brief Title: Observational Study of Botox® Treatment for Patients With Upper Limb Adult Spasticity
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/NS/SPA/018
Record Dates: First submitted 2011-06-30; First posted 2011-07-04 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2013-12

CONDITIONS: Muscle Spasticity
MeSH Terms: conditions — Muscle Spasticity | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- botulinum toxin Type A: Botulinum toxin Type A treatment at a dose determined by the physician at Baseline followed by a second botulinum toxin Type A treatment approximately 12 weeks later if applicable.
  Interventions: Biological: botulinum toxin Type A

INTERVENTIONS:
Biological: botulinum toxin Type A — Botulinum toxin Type A treatment at a dose determined by the physician at Baseline followed by a second botulinum toxin Type A treatment approximately 12 weeks later if applicable.
  Other Names: BOTOX®

SUMMARY:
This is a prospective, non-interventional, observational study to collect data on the use of botulinum toxin Type A in a routine setting in patients with upper limb adult spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with upper limb spasticity following a stroke
* Eligible to receive botulinum toxin Type A
* No previous botulinum toxin Type A therapy

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with upper limb spasticity following stroke who are eligible to receive botulinum toxin Type A treatment
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Itzehoe, Schleswig-Holstein, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin Type A
Started | 108
Completed | 100
Not Completed | 8
Not completed — Lost to Follow-up | 7
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 108
Age, Customized [Number; unit: Participants]
  18-30 Years | 8
  31-40 Years | 13
  41-50 Years | 22
  51-60 Years | 23
  61-70 Years | 24
  71-80 Years | 14
  81-90 Years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 61

OUTCOME MEASURES:

1. Primary Outcome: Muscle Tone as Measured by the Modified Ashworth Scale (MAS) in the Elbow at Baseline
Description: The MAS assessed the degree of muscle tone during movement of the elbow compared to normal muscle tone using a 6-point scale where: 0=no increase in muscle tone, 1=Slight increase in muscle tone manifested by a catch and release or by minimal resistance at the end of the range of motion when the part is moved, 1+=Slight increase in muscle tone manifested by a catch followed by minimal resistance throughout the remainder of the range of motion, 2=Marked increase in muscle tone through most of the range of motion but affected part easily moved, 3=Considerable increase in muscle tone passive movement difficult or 4=Affected part rigid in movement or extension. A low score indicated little or no stiffness (best). A high score indicated severe stiffness (worse). The number of participants in each score category is presented.
Time Frame: Baseline
Population: Efficacy population included all participants who received BOTOX® not previously treated with botulinum toxin.
Measure: Number; unit: Participants
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 101
Participants
  0=No Increase | 2
  1=Slight Increase | 6
  1+=Slight Increase | 18
  2=Marked Increase | 39
  3=Considerable Increase | 30
  4=Affected part rigid | 6

2. Primary Outcome: Muscle Tone as Measured by the Modified Ashworth Scale (MAS) in the Elbow at Week 24
Description: as for outcome 1
Time Frame: Week 24
Population: Participants from the Efficacy population (all participants who received BOTOX® not previously treated with botulinum toxin) who had data available for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 89
Participants
  0=No Increase | 2
  1=Slight Increase | 26
  1+=Slight Increase | 43
  2=Marked Increase | 12
  3=Considerable Increase | 5
  4=Affected part rigid | 1

3. Primary Outcome: Muscle Tone as Measured by the Modified Ashworth Scale (MAS) in the Wrist at Baseline
Description: The MAS assessed the degree of muscle tone during movement of the wrist compared to normal muscle tone using a 6-point scale where: 0=no increase in muscle tone, 1=Slight increase in muscle tone manifested by a catch and release or by minimal resistance at the end of the range of motion when the part is moved, 1+=Slight increase in muscle tone manifested by a catch followed by minimal resistance throughout the remainder of the range of motion, 2=Marked increase in muscle tone through most of the range of motion but affected part easily moved, 3=Considerable increase in muscle tone passive movement difficult or 4=Affected part rigid in movement or extension. A low score indicated little or no stiffness (best). A high score indicated severe stiffness (worse). The number of participants in each score category is presented.
Time Frame: Baseline
Population: Efficacy population included all participants who received BOTOX® not previously treated with botulinum toxin.
Measure: Number; unit: Participants
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 101
Participants
  0=No Increase | 3
  1=Slight Increase | 9
  1+=Slight Increase | 16
  2=Marked Increase | 29
  3=Considerable Increase | 35
  4=Affected part rigid | 9

4. Primary Outcome: Muscle Tone as Measured by the Modified Ashworth Scale (MAS) in the Wrist at Week 24
Description: as for outcome 3
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 89
Participants
  0=No Increase | 5
  1=Slight Increase | 31
  1+=Slight Increase | 31
  2=Marked Increase | 15
  3=Considerable Increase | 6
  4=Affected part rigid | 1

5. Primary Outcome: Muscle Tone as Measured by the Modified Ashworth Scale (MAS) in the Fingers at Baseline
Description: The MAS assessed the degree of muscle tone during movement of the fingers compared to normal muscle tone using a 6-point scale where: 0=no increase in muscle tone, 1=Slight increase in muscle tone manifested by a catch and release or by minimal resistance at the end of the range of motion when the part is moved, 1+=Slight increase in muscle tone manifested by a catch followed by minimal resistance throughout the remainder of the range of motion, 2=Marked increase in muscle tone through most of the range of motion but affected part easily moved, 3=Considerable increase in muscle tone passive movement difficult or 4=Affected part rigid in movement or extension. A low score indicated little or no stiffness (best). A high score indicated severe stiffness (worse). The number of participants in each score category is presented.
Time Frame: Baseline
Population: Efficacy population included all participants who received BOTOX® not previously treated with botulinum toxin.
Measure: Number; unit: Participants
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 101
Participants
  0=No Increase | 0
  1=Slight Increase | 5
  1+=Slight Increase | 15
  2=Marked Increase | 20
  3=Considerable Increase | 47
  4=Affected part rigid | 14

6. Primary Outcome: Muscle Tone as Measured by the Modified Ashworth Scale (MAS) in the Fingers at Week 24
Description: as for outcome 5
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 89
Participants
  0=No Increase | 4
  1=Slight Increase | 34
  1+=Slight Increase | 27
  2=Marked Increase | 17
  3=Considerable Increase | 5
  4=Affected part rigid | 2

7. Primary Outcome: Muscle Tone as Measured by the Modified Ashworth Scale (MAS) in the Thumb at Baseline
Description: The MAS assessed the degree of muscle tone during movement of the thumb compared to normal muscle tone using a 6-point scale where: 0=no increase in muscle tone, 1=Slight increase in muscle tone manifested by a catch and release or by minimal resistance at the end of the range of motion when the part is moved, 1+=Slight increase in muscle tone manifested by a catch followed by minimal resistance throughout the remainder of the range of motion, 2=Marked increase in muscle tone through most of the range of motion but affected part easily moved, 3=Considerable increase in muscle tone passive movement difficult or 4=Affected part rigid in movement or extension. A low score indicated little or no stiffness (best). A high score indicated severe stiffness (worse). The number of participants in each score category is presented.
Time Frame: Baseline
Population: Efficacy population included all participants who received BOTOX® not previously treated with botulinum toxin.
Measure: Number; unit: Participants
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 101
Participants
  0=No Increase | 1
  1=Slight Increase | 13
  1+=Slight Increase | 19
  2=Marked Increase | 19
  3=Considerable Increase | 36
  4=Affected part rigid | 13

8. Primary Outcome: Muscle Tone as Measured by the Modified Ashworth Scale (MAS) in the Thumb at Week 24
Description: as for outcome 7
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 89
Participants
  0=No Increase | 19
  1=Slight Increase | 29
  1+=Slight Increase | 18
  2=Marked Increase | 11
  3=Considerable Increase | 11
  4=Affected part rigid | 1

ADVERSE EVENTS:
Arm/Group | Botulinum Toxin Type A
Serious Adverse Events (participants affected / at risk) | 1/108
Other Adverse Events (participants affected / at risk) | 0/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (N=108)
Status epilepticus (Nervous system disorders) | 1
Bacteraemia (Infections and infestations) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Gastroenteritis norovirus (Gastrointestinal disorders) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Endocrine disorders) | 1
Hypoglycaemia (Endocrine disorders) | 1
Candiduria (Renal and urinary disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Death (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.